CLINICAL TRIAL: NCT04799457
Title: Comparison the Effect of Uterine Closure Technique Difference on Uterine Niche After Caesarean Delivery.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Ergul Demircivi Bor, Principal Investigator, Kanuni Sultan Suleyman Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2021/0077
Record Dates: First submitted 2021-03-05; First posted 2021-03-16 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Uterine Niche; Closure; Incomplete, Uterus
Keywords: niche; caesarean section; technique; uterine closure
MeSH Terms: interventions — Suture Techniques

STUDY DESIGN:
Intervention Model Description: Double Blinded Randomised Controlled Trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: One study control person is organizing the whole trial and provides blinding to both sides (participants and care provider).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Classical caesarean group (No Intervention): Care providers are applying standard caesarean procedure for participants.
- Study caesarean group (Experimental): Care providers are applying additional sutures to standard caesarean procedure for participants.
  Interventions: Other: Suture technique

INTERVENTIONS:
Other: Suture technique — We wil apply additional sutures to classical caesarean procedure.
  Arms: Study caesarean group

SUMMARY:
Caesarean section scar may have result as isthmocele or scar detachment during pregnancy which is in few years after previous delivery. Uterine niche is the most effectively used measurement side of uterus to estimate for these detachment complications. The aim of this study is to support this niche site by supporting the classical uterine closure technique.

DETAILED DESCRIPTION:
Cesarean delivery rate continues to increase in world in concern with uterine scar complications as placental invasion abnormalities, isthmocele or previous scar detachment during pregnancy (post surgical long term complications). Uterine niche is the presence of a hypoechoic area within the myometrium on the lower uterine segment, showing a defect of the myometrium at the site of a previous cesarean delivery. Some surgical techniques have been trying to support this area to prevent the post surgical long term complications. In this study the investigators have been trying to find out a new technique by applying supporting sutures during uterine closure in cesarean section. Three months after the surgery, the uterine niche measurement will be examined with ultrasonography for both study and classical groups and results will be compared between the groups.

ELIGIBILITY:
Inclusion Criteria:

* Primigravid elective caesarian delivery candidates
* The participants will have not any uterine contraction or cervical dilatation before delivery.
* Having no systemic or obstetric illnesses
* Participants who are accept to participate in this study with their written consent.

Exclusion Criteria:

* Previous caesarian delivery
* Having uterine contraction or cervical dilatation
* Smoking cigarettes
* Having systemic or obstetric illnesses

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — This trial will be conducted at an obstetrics and gynecology clinic.
Enrollment: 100 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants for each group for study | Up to 9 months
  We will try to reach fifty participants for each group (study group as classical cesarean with supporting suture and control group as classical cesarean) . When we reach to all participants we will stop to enroll the participants.

CONTACTS AND LOCATIONS:
Overall Officials: Ergul Demircivi Bor, Principal Investigator — Prof Dr Suleyman Yalcin Goztepe City Hospital
Locations (1):
- Prof Dr Suleyman Yalcin Goztepe City Hospital, Istanbul, Kadikoy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bennich G, Rudnicki M, Wilken-Jensen C, Lousen T, Lassen PD, Wojdemann K. Impact of adding a second layer to a single unlocked closure of a Cesarean uterine incision: randomized controlled trial. Ultrasound Obstet Gynecol. 2016 Apr;47(4):417-22. doi: 10.1002/uog.15792. PMID 26489989
- [Result] Roberge S, Demers S, Girard M, Vikhareva O, Markey S, Chaillet N, Moore L, Paris G, Bujold E. Impact of uterine closure on residual myometrial thickness after cesarean: a randomized controlled trial. Am J Obstet Gynecol. 2016 Apr;214(4):507.e1-507.e6. doi: 10.1016/j.ajog.2015.10.916. Epub 2015 Nov 11. PMID 26522861
- [Result] Sevket O, Ates S, Molla T, Ozkal F, Uysal O, Dansuk R. Hydrosonographic assessment of the effects of 2 different suturing techniques on healing of the uterine scar after cesarean delivery. Int J Gynaecol Obstet. 2014 Jun;125(3):219-22. doi: 10.1016/j.ijgo.2013.11.013. Epub 2014 Feb 28. PMID 24680843
- [Result] Stegwee SI, Jordans I, van der Voet LF, van de Ven PM, Ket J, Lambalk CB, de Groot C, Hehenkamp W, Huirne J. Uterine caesarean closure techniques affect ultrasound findings and maternal outcomes: a systematic review and meta-analysis. BJOG. 2018 Aug;125(9):1097-1108. doi: 10.1111/1471-0528.15048. Epub 2018 Jan 30. PMID 29215795